CLINICAL TRIAL: NCT04754412
Title: Writing to Heal: A Culturally Based Brief Expressive Writing Intervention for Chinese Immigrant Breast Cancer Survivors
Brief Title: Culturally Based Brief Expressive Writing Intervention for the Improvement of Health in Chinese Immigrant Stage 0-III Breast Cancer Survivors, Writing to Heal Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-0708; NCI-2020-14096 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0708 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage 0 Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Carcinoma In Situ | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (control writing) (Active Comparator): Patients write about facts regarding their cancer diagnosis and treatment for 3 weekly 30-minute sessions.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (self-regulation writing) (Experimental): Patients write about stress and coping, emotional disclosure, and benefit finding for 3 weekly 30-minute sessions.
  Interventions: Other: Behavioral, Psychological or Informational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (self-cultivation writing) (Experimental): Patients write about positive thoughts and feelings regarding their breast cancer experience for 3 weekly 30-minute sessions.
  Interventions: Other: Behavioral, Psychological or Informational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Behavioral, Psychological or Informational Intervention — Write about stress and coping, emotional disclosure, and benefit finding
  Arms: Arm II (self-regulation writing)
Other: Behavioral, Psychological or Informational Intervention — Write about positive thoughts and feelings regarding their breast cancer experience
  Arms: Arm III (self-cultivation writing)
Other: Best Practice — Write about facts regarding their cancer diagnosis and treatment
  Other Names: standard of care; standard therapy
  Arms: Arm I (control writing)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the effect of a culturally based brief expressive writing intervention in improving the health of Chinese immigrant stage 0-III breast cancer survivors. Culturally based brief expressive writing interventions may help researchers learn more about the experiences of Chinese immigrant breast cancer survivors and how writing about their experiences may affect their health.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the health benefits of expressive writing compared with the control condition.

II. To characterize how acculturation moderates the effects of expressive writing interventions.

III. To identify mechanisms explaining the benefits of the interventions using mixed methods.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I (CONTROL): Patients write about facts regarding their cancer diagnosis and treatment for 3 weekly 30-minute sessions.

ARM II (SELF-REGULATION): Patients write about stress and coping, emotional disclosure, and benefit finding for 3 weekly 30-minute sessions.

ARM III (SELF-CULTIVATION): Patients write about positive thoughts and feelings regarding their breast cancer experience for 3 weekly 30-minute sessions.

After completion of study, patients are followed up at 6 weeks and at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with stage 0-III breast cancer.
2. Completed primary treatment, including surgery, chemotherapy, radiation therapy, immune therapy, and/or targeted therapy within the preceding 5 years.
3. Foreign-born Chinese women (aged 18 and older) who lived in the U.S. for at least six months in the past.

Exclusion Criteria:

1. Exclusion criteria include inability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QOL) | Up to 12 months
  Quality of life will be measured by the Functional Assessment of Cancer Therapy for patients with breast cancer (FACT-B). The scale contains 27 items that assess perceived QoL in four domains: physical well-being, social well-being, emotional well-being and functional well-being. Items are rated on a 5-point scale from 0 - not at all, to 4 - very much. Total scores range between 0 and 108, with higher scores indicating better quality of life

SECONDARY OUTCOMES:
Perceived stress | Up to 12 months
  Perceived stress will be measured by the Perceived Stress Scale. The current perceived stress has 4 items. Participants rate the degree to which they perceive their life situation, as described in each item, using a five-point Likert scale from 0 - never, to 4 - very often. Total scores range between 0 and 40; higher scores indicate higher perceived stress.
Stress biomarker - alpha amylase | Up to 6 weeks
  Alpha amylase will be assessed via saliva samples. Higher levels of perceived stress are associated with dysregulated salivary alpha-amylase levels.
Stress biomarker-cortisol | Up to 6 weeks
  Salivary cortisol will be assessed via saliva samples. Higher levels of perceived stress are associated with dysregulated cortisol levels.
Number of medical appointments for cancer-related morbidities | Up to 12 months
  Will include appointments for non-routine cancer-related problems (e.g., lymphedema, breast symptoms, or possible recurrence) but exclude scheduled check-ups and non-routine medical appointments for other problems, such as flu symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Lu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Lu Q, Lun D, Dawkins-Moultin L, Li Y, Chen M, Giordano SH, Pennebaker JW, Young L, Wang C. Study protocol for writing to heal: A culturally based brief expressive writing intervention for Chinese immigrant breast cancer survivors. PLoS One. 2024 Sep 26;19(9):e0309138. doi: 10.1371/journal.pone.0309138. eCollection 2024. PMID 39325778
- See also: M D Anderson Cancer Center — http://www.mdanderson.org